CLINICAL TRIAL: NCT07141667
Title: Erector Spinae Plane Block Using Liposomal Bupivacaine Versus Bupivacaine Hydrochloride for Video-assisted Thoracic Surgery:Comparing Local Anesthetics on Quality of Recovery and Pain Score:A Randomised,Single-blind,Clinical Trial
Brief Title: Randomized Trial of Erector Spinae Plane Block Using Liposomal Bupivacaine Versus Bupivacaine Hydrochloride on Quality of Recovery for Video-assisted Thoracic Surgery
Acronym: LB-ESPB
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LY2025-199-A
Record Dates: First submitted 2025-07-21; First posted 2025-08-26 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Regional Anesthesia Morbidity; Pain, Postoperative
Keywords: quality of recovery; erector spinae plane block; liposomal bupivacaine; video-assisted thoracic surgery
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine

STUDY DESIGN:
Intervention Model Description: A single-blind, prospective, randomized controlled trial. Eligible patients scheduled for elective unilateral thoracic pulmonary resection will be randomly allocated to either the liposomal bupivacaine group or the bupivacaine HCL group. Patients in the liposomal bupivacaine group will undergo ultrasound-guided erector spinae plane block with liposomal bupivacaine, whereas those in the bupivacaine HCL group will receive ultrasound-guided erector spinae plane nerve block with bupivacaine hydrochloride.
Who Masked: Participant, Outcomes Assessor
Masking Description: This study adopts a single-blind design, where participants will be kept blinded to their assigned groups to minimize bias in subjective evaluations. Anesthesia providers will be responsible for screening and enrolling eligible patients, as well as administering the assigned anesthesia protocols. Importantly, the roles of anesthesia providers and postoperative follow-up personnel will be strictly separated, with the latter remaining unaware of the randomization details throughout the entire study period.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bupivacaine HCL Group (Active Comparator): Erector spinae plane block with normal saline 10ml and bupivacaine HCL 0.5% 20ml
  Interventions: Procedure: Erector spinae plane block with bupivacaine HCL
- Liposomal Bupivacaine Group (Experimental): Erector spinae plane block with normal saline 10ml and liposomal bupivacaine 1.33% 20ml
  Interventions: Procedure: Erector spinae plane block with liposomal bupivacaine

INTERVENTIONS:
Procedure: Erector spinae plane block with liposomal bupivacaine — In the anesthesia induction suite, the anesthesiologist administers an ultrasound-guided erector spinae plane (ESP) block under local anesthesia prior to the induction of general anesthesia. The procedure involves the sequential injection of 10 mL of normal saline, followed by the administration of 20 mL of 1.33% liposomal bupivacaine.
  Arms: Liposomal Bupivacaine Group
Procedure: Erector spinae plane block with bupivacaine HCL — In the anesthesia induction suite, the anesthesiologist administers an ultrasound-guided erector spinae plane (ESP) block under local anesthesia prior to the induction of general anesthesia. The procedure involves the sequential injection of 10 mL of normal saline, followed by the administration of 20 mL of 0.5% bupivacaine HCL.
  Arms: Bupivacaine HCL Group

SUMMARY:
Video-assisted thoracoscopic surgery (VATS) has emerged as the standard surgical modality for pulmonary tumor. Compared with open thoracotomy, VATS is associated with reduced surgical trauma, attenuated postoperative pain, and a lower incidence of postoperative pulmonary complications. Nevertheless, 27-63% of VATS patients still develop moderate to severe postoperative pain, with the incidence of chronic postsurgical pain (CPSP) remaining at 25-44%.

Regional analgesic techniques constitute a pivotal component of enhanced recovery after surgery (ERAS) protocols in thoracic surgery. Thoracic epidural analgesia (TEA) and paravertebral block (PVB) have been regarded as the gold-standard regional analgesic modalities for open thoracotomy. Accumulating evidence indicates that erector spinae plane block (ESPB) achieves postoperative analgesic efficacy comparable to that of PVB. In contrast to TEA, both PVB and ESPB are associated with a lower risk of complications such as hypotension, urinary retention, and epidural hematoma.

A recent randomized controlled trial comparing continuous ESPB and continuous PVB demonstrated that continuous ESPB improves the quality of postoperative recovery in VATS patients. Previous studies have also confirmed that single-injection ESPB provides superior recovery quality and analgesic efficacy compared with single-injection PVB in VATS patients. However, single-dose nerve block only exert effects for 8-12 hours, while continuous nerve blocks may increase the risk of infection and compromise patient comfort. Moderate to severe postoperative pain in VATS patients predominantly occurs within the first 48 hours postoperatively, with the most intense pain typically observed on the first postoperative day. Therefore, there is an urgent need to explore analgesic techniques with prolonged duration and fewer complications for application in VATS.

Liposomal bupivacaine, a novel extended-release local anesthetic approved by the FDA for clinical use, can prolong the duration of local anesthesia to 72 hours. Its clinical efficacy in procedures such as brachial plexus block has been validated. However, the application of liposomal bupivacaine in erector spinae plane block for VATS, and its impact on the quality of postoperative recovery, remains unreported.This study will test the hypothesis that erector spinae plane block with liposomal bupivacaine for VATS can enhance patients' quality of recovery-15 score (QoR-15) at 48 h.

DETAILED DESCRIPTION:
This is a prospective randomized controlled trial. Patients scheduled for elective video-assisted thoracoscopic pulmonary resection will be randomly assigned to two groups: the liposomal bupivacaine group, which will undergo erector spinae plane block with liposomal bupivacaine, and the bupivacaine hydrochloride group, which will receive erector spinae plane block with bupivacaine hydrochloride. Quality of recovery-15 score (QoR-15) and other outcome measures will be observed, and our hypothesis is that erector spinae plane block with liposomal bupivacaine can enhance patients' quality of recovery-15 score (QoR-15) at 48 h.

In the anesthesia induction suite, the anesthesiologist administers an ultrasound-guided erector spinae plane (ESP) block prior to the induction of general anesthesia. The procedure involves the sequential injection of 10 mL of normal saline, followed by the administration of 0.5% bupivacaine HCL 20ml or 1.33% liposomal bupivacaine 20ml.

Postoperatively, the following analgesic protocols are administered routinely:

Basic analgesia: Parecoxib sodium (a non-steroidal anti-inflammatory drug) 40 mg, every 12 hours;Patient-controlled intravenous analgesia (PCIA): A background infusion of sufentanil at 2 μg/h, with patient-controlled analgesia (PCA) boluses of sufentanil 2 μg and a lockout period of 15 minutes;Postoperative rescue analgesia: If NRS score is ≥ 4, the attending physician will administer rescue analgesia, which will be documented in the medical record.

Safety reporting: Any unexpected complications that may arise from this trial will be documented and reported to the principal investigator and the relevant hospital patient safety board.

Sample size and justification: The primary outcome will be the QoR-15 score at 48 hours post operatively.According to published studies on quality of recovery, the minimal clinically important difference (MCID) for the QoR-15 score after surgery is 8. For major surgeries, the standard deviation (SD) of postoperative QoR-15 scores typically ranges from 10 to 16, and an SD of 12 was selected for this study. Using a two-tailed test with a significance level of α=0.05 and a test power of 1-β=0.8, the sample size calculated for each group (for comparison between the two groups) was 36 participants. With an estimated dropout rate of 10%, the final sample size was determined to be 40 participants per group, resulting in a total sample size of 80 participants.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 yr of age
* ASA physical status 1 to 3
* Undergoing unilateral lung VATS under general anesthesia
* Obtaining informed consent from patients or legal representative

Exclusion Criteria:

* Unexpected convention of VATS to open thoracotomy,or unexpected post-operative admission to ICU for continued ventilation
* Unable to understand the Quality of Recovery-15 (QoR-15) and Numerical Rating Scale(NRS)
* Allergy to or contraindications for amide local anesthetics,opioids,or NSAIDs
* Long-term treatment with opioids or corticosteroids (>2 weeks)
* Drug use or substance abuse within the past 2 years
* Consuming more than 3 standard drinks per day (10g of alcohol,equivalent to 50g of Chinese high-alcohol liquor)
* Pre existing dementia that may interfere with perioperative assessment
* Contraindications for nerve block,including infection or tumor at the puncture site,definitively diagnosed diabetic peripheral neuropathy
* Suffering from severe hepatic insufficiency (Child-Pugh C),or severe renal insufficiency with dialysis,or severe heart failure (METS<4)
* Pregnant or lactating women
* Previous thoracic surgeries (such an thoracic surgery or breast surgery),or preoperatively pathological pain conditions (e.g.,metastatic tumors,herpes zoster,etc)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2028-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Quality of recovery-15 score (QoR-15) at 48 h | 48 hours postoperative
  QoR-15 is a 15-parameter questionnaire which has been recommended as an optimum tool to evaluate overall patient recovery after surgery and this includes postoperative pain. Participants will complete this questionnaire at 48 hours after their surgery. It is scored between 0 and 150, where 150 indicates that the patient has had an excellent recovery.

SECONDARY OUTCOMES:
Quality of recovery-15 score (QoR-15) at 24 h | 24 hours postoperative
  QoR-15 is a 15-parameter questionnaire which has been recommended as an optimum tool to evaluate overall patient recovery after surgery and this includes postoperative pain. Participants will complete this questionnaire at 48 hours after their surgery. It is scored between 0 and 150, where 150 indicates that the patient has had an excellent recovery.
Numerical Rating Scale (NRS) for pain at rest when leaving the PACU, as well as at 4 hours, 24 hours, and 48 hours postoperatively | Upon discharge from the recovery room(PACU),4 hours,24 hours and 48 hours postoperative
  Numerical Rating Scale pain score is measured from 0 to 10 where 0 is no pain and 10 is severe pain.
Numerical Rating Scale (NRS) for pain during coughing when leaving the PACU, as well as at 4 hours, 24 hours, and 48 hours postoperatively | Upon discharge from the recovery room(PACU),4 hours,24 hours and 48 hours postoperative
  Numerical Rating Scale pain score is measured from 0 to 10 where 0 is no pain and 10 is severe pain.
Area under the curve (AUC) of NRS for pain at rest and during coughing within 48 hours | 48 hours postoperative
  Numerical Rating Scale pain score is measured from 0 to 10 where 0 is no pain and 10 is severe pain.
Cumulative consumption of opioids within 48 hours postoperatively | 48 hours postoperative
  Dose of opioids consumed (in morphine equivalents) by participants
Incidence of pruritus and incidence of nausea and vomiting within 48 hours postoperatively | 48 hours postoperative
  The incidence of postoperative pruritus is the proportion of patients who experience pruritus; the incidence of postoperative nausea and vomiting is the proportion of patients who experience nausea and vomiting.Incidence of nausea and vomiting will be defined as any nausea, emetic episodes (vomiting or retching), or both.Nausea is diagnosed when the patient has gastrointestinal symptoms but does not vomit stomach contents. Vomiting is diagnosed when the patient has gastrointestinal symptoms and retching or vomits gastric contents. Retching refers to the act of vomiting, but no stomach contents are vomited out.
Overall Benefit of Analgesia Score (OBAS) at 48 hours postoperatively | 48 hours postoperative
  The Overall Benefit of Analgesia Score (OBAS) is a multi-dimensional survey that measures a patient's benefit from postoperative pain therapy. It assesses pain intensity, opioid-related adverse events, and patient satisfaction with analgesia. Each of 7 questions are scored on a scale from 0 to 4 where 0=minimal/not at all and 4=maximum/very much. Total scores range from 0 to 28 with lower scores representing greater benefit from analgesic therapy.